CLINICAL TRIAL: NCT06825559
Title: A Phase 1, Open-label, Single Arm Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Saroglitazar Magnesium Dosed on Alternate Days in Subjects Having Moderate Hepatic Impairment With Cirrhosis Due to Cholestatic Liver Disease
Brief Title: Evaluate PK & Safety of Saroglitazar in Subjects With Moderate Hepatic Impairment Due to Cholestatic Liver Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARO.24.003
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cholestatic Liver Disease
Keywords: Saroglitazar Magnesium; Primary Biliary Cholangitis; PBC; Pharmacokinetics
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — saroglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Saroglitazar Magnesium 1 mg (Experimental): Saroglitazar Magnesium 1 mg tablet orally administered on alternate days in the morning before breakfast without food, for the duration of treatment (29 days)
  Interventions: Drug: Saroglitazar Magnesium 1 mg

INTERVENTIONS:
Drug: Saroglitazar Magnesium 1 mg — Saroglitazar Magnesium 1 mg will be assigned to all participants enrolled in this open label study
  Other Names: Not any

SUMMARY:
Evaluating Pharmacokinetic and safety of Saroglitazar Magnesium 1 mg when dosed on alternate days in subjects having moderate hepatic impairment with cirrhosis due to cholestatic liver disease

DETAILED DESCRIPTION:
A phase 1, open-label, single arm study to evaluate pharmacokinetics, safety, and tolerability of Saroglitazar Magnesium dosed on alternate days in subjects having moderate hepatic impairment with cirrhosis due to cholestatic liver disease

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female aged 18 to 80 years (both inclusive) at the time of signing the ICF.
2. Body mass index within the range 18.0 to 48.0 kg/m2 (inclusive) at screening.
3. Ability to swallow and retain oral medication.
4. Subjects having documented history of hepatic impairment with cirrhosis due to cholestatic liver disease having Child-Pugh Turcotte score 7 to 9. If the hepatic impairment classification for the subject is not the same at screening and Day -1, enrolment of the subject into a hepatic category group will be at the discretion of the investigator.
5. Laboratory test values must be clinically acceptable to the investigator and meet all the following parameters at screening:

   Alkaline Phosphatase > upper limit of normal Alanine aminotransferase/Aspartate aminotransferase value ≤ 10 × upper limit of normal Absolute neutrophil count ≥ 750/mm3 Platelets ≥ 25,000/mm3 Hemoglobin ≥ 8 g/dL α-fetoprotein <50 ng/mL or 50-80 ng/mL with negative imaging study (Ultrasound [US], computed tomography scan [CT], Magnetic Resonance Imaging [MRI]). Imaging study that excluded presence of liver cancer (US in the preceding 6 months and CT or MRI in the preceding 1 year)
6. Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

1. Any significant or unstable medical condition or other instability that would prevent the subject from participating in the study as determined by the investigator
2. History of malignancy of any type in the last 3 years of screening, with the exception of the following: in situ cervical or breast cancer or surgically excised non-melanoma skin cancers (i.e., basal cell or squamous cell carcinoma).
3. History of stomach or intestinal surgery or resection within 6 months of screening that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair will be allowed).
4. The history of any significant drug allergy (such as anaphylaxis) deemed clinically relevant by the investigator.
5. Any major surgery within 3 months of screening.
6. Donation of blood or blood products within 3 months of screening.
7. Active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment or symptoms of active infectious disease within 2 weeks of screening.
8. Receiving or has received any investigational drug within 30 days or 5 half-lives (whichever is longer), before receiving Saroglitazar Magnesium.
9. Estimated glomerular filtration rate (<45 mL/min/1.73 m2 by CKD-EPI 2021 formula at screening.
10. Any individual with poor peripheral venous access.
11. Receipt of blood products within 1 month of check in.
12. Human immunodeficiency virus type 1 antibody positive at screening.
13. Other known causes of liver disease, such as non-alcoholic steatohepatitis , alcoholic steatohepatitis, autoimmune hepatitis, or acute or chronic viral hepatitis (including Hepatitis B and C) as determined by the investigator and subject's medical records.
14. Subjects who have had a change in hepatic disease status within 30 days of screening, as documented by the subject's medical history and deemed clinically significant by the investigator.
15. Subjects having - History of gastrointestinal bleeding within 1 month of screening. Current functioning organ transplant. Evidence of severe ascites requiring frequent paracentesis in the opinion of the investigator.
16. Pregnancy-related exclusions, including:

Pregnant/lactating female (including positive pregnancy test at screening) Pregnancy should be avoided by male and female subjects either by true abstinence or the use of an acceptable effective contraceptive measures for the duration of the study and for at least 1 month after the end of the study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of Saroglitazar: Cmax | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  Maximum plasma concentration (Cmax)
Pharmacokinetics of Saroglitazar: Tmax | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  Time to reach maximum plasma concentration (Tmax)
Pharmacokinetics of Saroglitazar: AUCt | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve till the last time point
Pharmacokinetics of Saroglitazar: AUCi | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve extrapolated to the infinity
Pharmacokinetics of Saroglitazar: Kel | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The elimination rate constant
Pharmacokinetics of Saroglitazar: AUCtau | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve in a 48 hours dosing interval
Pharmacokinetics of Saroglitazar: t1/2 | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The elimination half-life
Pharmacokinetics of Saroglitazar: Vd/F | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The apparent volume of distribution
Pharmacokinetics of Saroglitazar: CL/F | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The apparent clearance

SECONDARY OUTCOMES:
Number of participants with adverse events [Safety and Tolerability] | From baseline to End of study (35 days)
  Number of participants with adverse events
Pharmacokinetics of Saroglitazar sulfoxide: Tmax | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  Time to reach maximum plasma concentration
Pharmacokinetics of Saroglitazar sulfoxide: Cmax | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  Maximum plasma concentration
Pharmacokinetics of Saroglitazar sulfoxide: CL/F | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The apparent clearance
Pharmacokinetics of Saroglitazar sulfoxide: Vd/F | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The apparent volume of distribution
Pharmacokinetics of Saroglitazar sulfoxide: t1/2 | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The elimination half-life
Pharmacokinetics of Saroglitazar sulfoxide: AUCtau | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve in a 48 hours dosing interval
Pharmacokinetics of Saroglitazar sulfoxide: Kel | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The elimination rate constant
Pharmacokinetics of Saroglitazar sulfoxide: AUCi | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve extrapolated to the infinity
Pharmacokinetics of Saroglitazar sulfoxide: AUCt | PK sampling timepoints: pre- dose, 20 min, 40 min, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36, and 48 hours post-dose of Day 1 and Day 29
  The area under plasma concentration vs. time curve extrapolated to the infinity
Change from baseline in alkaline phosphatase levels | From baseline to end of treatment (29 days)

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, Study Director — Zydus Therapeutics Inc.
Locations (1):
- Zydus Site US001, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Rodney P, Starzomski R. Constraints on the moral agency of nurses. Rhinology. 1993 Oct;69(9):23-6. No abstract available. PMID 11652809